CLINICAL TRIAL: NCT04821557
Title: Effect of Microbial Protease Supplementation on Postprandial Amino Acid Levels in Healthy Adults
Brief Title: Effect of Microbial Protease Supplementation on Postprandial Amino Acid Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: BIO-CAT, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21545
Record Dates: First submitted 2021-03-22; First posted 2021-03-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Protein Metabolism
Keywords: Protein; Amino Acids; Branched Chain Amino Acids; Leucine; Postprandial
MeSH Terms: interventions — Peptide Hydrolases; Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplement and placebo powders will be provided to the clinic in blindly coded containers. The code was generated by parties not responsible for data collection, analysis, or interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbial Protease Supplement (Experimental): A microbial protease supplement (31,875 Hemoglobin Unit Tyrosine base (HUT); protease activity) is taken with a 25g pea protein beverage. The test article will be provided in 250mg capsule form. Capsules will be opened and mixed into protein shake 5 minutes before ingestion.
  Interventions: Dietary Supplement: Protease + Protein
- Placebo (Maltodextrin) (Placebo Comparator): The placebo (maltodextrin) article will be provided in 250mg capsule form. Capsules will be opened and mixed into 25g pea protein shake 5 minutes before ingestion.
  Interventions: Dietary Supplement: Placebo + Protein

INTERVENTIONS:
Dietary Supplement: Protease + Protein — Participant will consume a microbial protease supplement (31,875 Hemoglobin Unit Tyrosine base (HUT); protease activity) combined with a pea protein beverage (25 g pea protein; Roquette Nutralys® S85F)
  Arms: Microbial Protease Supplement
Dietary Supplement: Placebo + Protein — Participant will consume a placebo supplement (250 mg maltodextrin) combined with a pea protein beverage (25 g pea protein; Roquette Nutralys® S85F)
  Arms: Placebo (Maltodextrin)

SUMMARY:
Dietary protein is digested in the stomach and intestines to smaller peptides and 20 individual amino acids which, when absorbed by the gut into circulation and taken up by skeletal muscle, help stimulate muscle protein synthesis (MPS). Amino acids also provide the building blocks for muscle proteins that contribute to lean mass gains and increased strength following resistance exercise. Therefore, strategies to efficiently maximize amino acid exposure without overconsumption are warranted.

Oral enzyme supplementation is a candidate approach to optimize amino acid absorption from dietary protein and protein supplements. Microbial proteases, approved for dietary supplement use, can theoretically speed up the conversion of protein and peptides to amino acids. Protease supplements have been marketed to promote muscle strength by optimizing amino acid absorption, however the clinical evidence is limited. This work will support that ingestion of protease supplements with a meal can allow individuals to more efficiently increase amino acid levels from a given amount of dietary protein.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 - 50 years
* Body mass index = 18.0-29.9 kg∙m-2

Exclusion Criteria:

* Age outside of range (20 - 50 y)
* Pregnancy
* Subject states they regularly consume probiotic supplements and are unwilling to stop at least one week prior to screening and throughout the study (Supplemental probiotics may include standalone probiotic supplements, vitamins with probiotics, and any foods supplemented with probiotics)
* Subject states they regularly consume supplemental enzymes and are unwilling to stop at least one week prior to screening and throughout the study (Supplemental enzymes may include standalone enzyme supplements, probiotic supplements with enzymes, and any medications containing enzymes)
* Abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
* Diabetes (fasting glucose ≥ 126 mg/dL)
* Active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix
* Liver failure (decompensated chronic liver disease)
* History of a significant cardiovascular event (e.g., myocardial infarction, heart failure, or stroke) ≤ 3 months prior to the screening visit
* Subject reports having undergone major surgery less than 6 weeks prior to enrollment in the study, or subject has planned inpatient surgery requiring 2 or more days of hospitalization during the entire study
* Currently being prescribed (by primary care physician or other health professional) medication or using an over the counter product that in the opinion of the study physician will have an effect on food digestion or nutrient absorption during the study (e.g., prescription orlistat [Xenical], over the counter orlistat [Alli])
* Alcohol intake an average of 3 or more servings per day (a serving defined as 4 oz wine, 12 oz beer, 1 oz spirits)
* Subject is deemed unsuitable for study based upon study physician assessment
* Irregular menstrual cycles
* Participation in other ongoing research that interferes with this study (e.g., conflicting diet, activity interventions, etc.)
* Any hospitalization or surgery for a metabolic, cardiovascular, or neuromusculoskeletal complication within the past year
* Allergy or hypersensitivity to latex or adhesives (bandages, medical tape, etc.)
* Chronic or frequent dizziness/fainting, and arm or leg weakness/numbness
* Mental Illness
* Hepatorenal, cardiovascular musculoskeletal, autoimmune, or neurological disease or disorder
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, non-steroidal anti-inflammatories, or acne medication)
* Unwillingness to comply with study procedures
* Weight unstable (variation >5% of bodyweight in last 6 months)
* Current or previous tobacco or marijuana use within the last 6 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Total plasma branched chain amino acid(BCAA) area under the curve(AUC) | Five-hours postprandial
  Five-hour area under the curve plasma levels of total BCAA following a protein shake tolerance test, change from baseline
  Free leucine, isoleucine, and valine (combined)
Plasma BCAA time-to-peak | Five-hours postprandial
  Time to peak plasma levels of total BCAA following a protein shake tolerance test, change from baseline
  Total of free leucine, isoleucine, and valine (combined)
Plasma BCAA C(MAX) | Five-hours postprandial
  C(MAX) plasma levels of total BCAA levels following a protein shake tolerance test, change from baseline
  Total of free leucine, isoleucine, and valine (combined)

SECONDARY OUTCOMES:
Plasma essential amino acid (EAA) AUC | Five-hours postprandial
  Five-hour area under the curve plasma levels of total EAA following a protein shake tolerance test, change from baseline
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan
Plasma Leucine AUC | Five-hours postprandial
  Five-hour area under the curve plasma levels of total EAA following a protein shake tolerance test, change from baseline
  Free leucine
Plasma Total amino acid (AA) AUC | Five-hours postprandial
  Five-hour area under the curve plasma levels of total AA following a protein shake tolerance test, change from baseline
  Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline
Plasma Insulin AUC | Five-hours postprandial
  Five-hour AUC plasma insulin following a protein shake tolerance test, change from baseline
Postprandial appetite, hunger, desire-to-eat | Five-hours postprandial
  Visual analog scale questionnaires designed to assess appetite, hunger, desire to eat, administered hourly. Scales from 0 - 100mm. Higher scores indicate higher appetite, hunger or desire to eat.
Gastrointestinal comfort | Five-hours postprandial
  Questionnaire (Y/N questions) to determine presence/absence of gastrointestinal discomfort, pain, bloating, and nausea.

OTHER OUTCOMES:
Plasma Glucose AUC | Five-hours postprandial
  <safety outcome> Five-hour AUC plasma glucose following a protein shake tolerance test, change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall; University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paulussen KJM, Askow AT, Deutz MT, McKenna CF, Garvey SM, Guice JL, Kesler RM, Barnes TM, Tinker KM, Paluska SA, Ulanov AV, Bauer LL, Dilger RN, Burd NA. Acute Microbial Protease Supplementation Increases Net Postprandial Plasma Amino Acid Concentrations After Pea Protein Ingestion in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled Trial. J Nutr. 2024 May;154(5):1549-1560. doi: 10.1016/j.tjnut.2024.03.009. Epub 2024 Mar 11. PMID 38467279